CLINICAL TRIAL: NCT06573450
Title: Preliminary Application and Evaluation of Exhaled Breath Condensate Biomarkers in Combined Allergic Rhinitis and Asthma Syndrome (CARAS)
Brief Title: Exhaled Breath Condensate Biomarkers in CARAS
Status: Recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EBC biomarkers in CARAS
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Combined Allergic Rhinitis and Asthma Syndrome
Keywords: CARAS; EBC; Biomarkers; Combination of disease and evidence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- acute exacerbation CARAS: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- chronic persistence CARAS: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- clinical control CARAS: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- acute exacerbation BA: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- chronic persistence BA: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- clinical control BA: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- intermittent AR: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- persistent AR: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey
- healthy individuals: Thirty subjects were included. No intervention was performed and only relevant patient information, blood and exhaled breath condensate were collected.
  Interventions: Other: questionnaire survey

INTERVENTIONS:
Other: questionnaire survey — subjects fill out questionnaires

SUMMARY:
To explore the differences in the expression of biomarkers in different sample types between the healthy population and different subgroups of the disease, and to screen for potential biomarkers in a more simple, direct and objective way. To screen the biomarkers that can be identified by CARAS Chinese medicine symptoms and different stages, and to provide a reference basis for individualised diagnosis and treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AR, BA and CARAS who meet the Western medical diagnostic criteria;
* Chinese medical evidence consistent with lung qi deficiency evidence, phlegm-heat congestion of the lung evidence, or wind-heat offending the lung evidence;
* Age 18 to 80 years;
* Voluntarily accepted the study and signed an informed consent form;
* Not participated in other clinical studies within 1 month before enrollment.

Exclusion Criteria:

* Patients with combined vasomotor rhinitis and eosinophilic non-allergic rhinitis, other non-allergic rhinitis diseases that can cause symptoms such as nasal congestion and runny nose;
* Patients who are participating in other drug trials;
* Patients with a combination of other serious systemic diseases;
* Pregnant or lactating women;
* Patients with confusion, disorders of consciousness, dementia, and various psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Allergic rhinitis (AR) is a common chronic inflammatory disease of the upper respiratory tract with paroxysmal sneezing, nasal congestion, watery nasal discharge and nasal itching as the main clinical symptoms. Bronchial asthma (BA) is a complex heterogeneous chronic inflammatory disease of the bronchi with recurrent symptoms of wheezing, shortness of breath, chest tightness, and coughing.AR usually coexists with BA, and about 70-90% of patients with asthma develop rhinitis, and about 40% of patients with rhinitis develop asthma. When AR and BA occur together, it is called combined allergic rhinitis and asthma syndrome (CARAS).
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Interleukin-2、4、5、13 (IL-2、4、5、13) | Basline
  Airway inflammation will be assessed using the IL-2、4、5、13.
Interferon-γ (IFN-γ) | Basline
  Airway inflammation will be assessed using the IFN-γ.
Tumor necrosis factor-β (TNF-β) | Basline
  Airway inflammation will be assessed using the TNF-β.
Eosinophil cationic proteins (ECP) | Basline
  Airway inflammation will be assessed using the ECP.
Immunoglobulin E (IgE) | Basline
  Airway inflammation will be assessed using the IgE.

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide (FeNO) | Basline
  Higher FeNO values indicate higher airway inflammation.
Forced expiratory volume in one second (FEV1) | Basline
  Lung function will be assessed using the FEV1.
Forced vital capacity (FVC) | Basline
  Lung function will be assessed using the FEV1.
FVC as the percentage of the predicted value (FVC%) | Basline
  Lung function will be assessed using the FVC%.
Forced expiratory volume in one second / forced vital capacity (FEV1/FVC) | Basline
  Lung function will be assessed using the FEV1/FVC.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Henan, Zhengzhou, China